CLINICAL TRIAL: NCT06822010
Title: A Phase II Trial of SeqUential GeMcitabine and MITomycin Treatment for Favorable High-Risk Upper Urinary Tract Urothelial Carcinoma (SUMMIT)
Brief Title: SeqUential GeMcitabine and MITomycin Treatment for Favorable High-Risk Upper Urinary Tract Urothelial Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Vignesh Packiam, Associate Professor, Rutgers, The State University of New Jersey
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 082411; Pro2024002505 (Other: Rutgers)
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-11

CONDITIONS: Urinary Bladder Cancer; Upper Tract Urothelial Cancer; Urothelial Cancer
Keywords: upper tract urothelial cancer; urothelial cancer; gemcitabine; jelmyto; mitomycin
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Gemcitabine

STUDY DESIGN:
Intervention Model Description: The study uses a Single Group Assignment model, where all participants enrolled in the trial will receive the same experimental intervention: sequential administration of gemcitabine and Jelmyto (mitomycin). The intervention is delivered directly into the kidney through a nephrostomy tube over six weekly treatments, with possible additional cycles based on the tumor's response.
  The objective of this model is to evaluate how this combination treatment affects tumor response, recurrence rates, and kidney preservation outcomes in participants with favorable high-grade upper tract urothelial carcinoma (UTUC). No control group or randomization is used, as the primary purpose is to determine the safety and efficacy of the sequential chemotherapy treatment in a focused patient population.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sequential Gemcitabine and Jelmyto Treatment (Gem/Jel) (Experimental): Participants in this arm will receive six weekly doses of sequential gemcitabine and Jelmyto (mitomycin) directly administered into the affected kidney through a nephrostomy tube. Depending on the tumor's response, participants may receive an additional six weekly doses or transition to a standard of care maintenance regimen. The primary goal of this arm is to evaluate the complete response rate, safety, and long-term outcomes such as recurrence-free survival and kidney preservation.
  Interventions:
  Drug: Gemcitabine (endoluminal administration)
  Drug: Jelmyto (gel-based mitomycin, endoluminal administration)
  Interventions: Drug: Sequential Gemcitabine and Jelmyto Treatment (Gem/Jel)

INTERVENTIONS:
Drug: Sequential Gemcitabine and Jelmyto Treatment (Gem/Jel) — Drug: Gemcitabine (endoluminal administration)
  Drug: Jelmyto (gel-based mitomycin, endoluminal administration)
  Other Names: Gemcitabine (endoluminal administration); Jelmyto (gel-based mitomycin, endoluminal administration)

SUMMARY:
This Phase II clinical trial, titled "A Phase II Trial of Sequential Gemcitabine and Mitomycin Treatment for Favorable High-Risk Upper Urinary Tract Urothelial Carcinoma (SUMMIT)," aims to evaluate the safety and effectiveness of a combination chemotherapy treatment for patients with favorable papillary high-grade upper tract urothelial carcinoma (UTUC). The study focuses on sequential administration of two drugs, gemcitabine and Jelmyto (a gel-based form of mitomycin), to potentially preserve kidney function and avoid nephroureterectomy (kidney removal), which is the current standard of care for participants with non-endoscopically resectable tumors.

DETAILED DESCRIPTION:
Participants enrolled in the study will receive six weekly doses of gemcitabine and Jelmyto delivered directly into the affected kidney through a nephrostomy tube. Based on the tumor's response, patients may receive an additional six doses or transition to a standard maintenance regimen. The primary goal is to assess the complete response rate of this treatment and determine its effectiveness in preserving kidney function while managing cancer recurrence. Secondary objectives include evaluating safety, recurrence-free survival at 12 and 24 months, and patient-reported outcomes over time.

The study is expected to last approximately 3 years, with participants undergoing regular follow-up evaluations. If the treatment is ineffective, standard procedures such as nephroureterectomy may still be performed.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following applicable inclusion criteria to participate in the study:

  1. Patient has signed Informed Consent Form and is willing and able to comply with all requirements of the protocol.
  2. Patient is at least 18 years of age.
  3. Naive or recurrent patients with High Grade Ta +/- CIS, non-invasive UTUC in the upper tract (pyelocalyceal system or ureter).
* Histologic confirmation with biopsy is necessary.
* All patients must undergo ureteroscopy with biopsy.
* Non-Invasive Papillary Carcinoma (HGTa) lesions must be maximally ablated with ≤ 15 mm residual papillary disease in total.

  4. Favorable high-grade upper tract urothelial carcinoma (UTUC) as per American Urological Association (AUA) risk stratification below (except that multifocality, obstruction, ureteral involvement, bladder involvement will be allowed).
  1. If the bladder is involved with NMIBC it should be treated prior to or during Gem/Jel treatments.

     5. Patients with ECOG (Eastern Cooperative Oncology Group) performance status <3 (with Karnofsky >40).

     6. Patients with life expectancy greater than 24 months at time of screening. 7. Patient has no active urinary tract infection (UTI) as confirmed by urine culture or urinalysis*.

     8. Female Patients of childbearing potential**, must have a negative serum pregnancy test at screening and must agree to use two acceptable & effective methods of contraception***, until 6 months post treatment 9. All sexually active male patients must agree to use a condom during intercourse, for at least 48 hours post each instillation.

     10. Male patients who have a partner that is a female of childbearing potential must agree to use two acceptable & effective methods of contraception until 6 months post treatment.

     11. Patients must not have any other medical condition(s) that make(s) their participation in the study unadvisable in the opinion of the investigator.

     Exclusion Criteria:

     Invasive upper tract urothelial carcinoma (suspected cT2-4 on imaging) or lymphadenopathy (cN1-3) Bilateral disease Patient is actively being treated or intends to be treated with systemic chemotherapy during the duration of the trial.

     4. Any other malignancy diagnosed within 2 years of trial entry with the exception of:

  a. Basal or squamous cell skin cancers, or b. Noninvasive cancer of the cervix, or c. Any other cancer deemed to be of low-risk for progression or patient morbidity during trial period (basal or squamous cell skin cancers, noninvasive cancer of the cervix, prostate cancer under active surveillance, renal cancer under active surveillance).

  4. Administration not feasible via nephrostomy tube. 5. Inability to deliver the investigational drug to the pyelocalyceal system. 6. Patient has any other medical or mental condition(s) that make(s) his/her participation in the trial unadvisable in the opinion of the treating urologist.

  7. Patient has contraindication to mitomycin C (MMC )treatment, or known sensitivity to MMC.

  8. Patient has an intractable bleeding disorder (e.g., coagulation factors deficiencies, Von Willebrand Disease).

  9. Patient is currently receiving any other investigational agents or has participated in a research protocol involving administration of an investigational product within the past 30 days prior to Visit 1.

  10. Pregnant (positive serum pregnancy test), planning to become pregnant during the trial period, breast-feeding, or of childbearing potential and not practicing reliable contraception***.

  * In case of a symptomatic UTI the patient will be treated with a full course of antibiotics, and the instillation will be postponed until resolution. In the case of asymptomatic bacteriuria, the use of prophylactic antibiotics and postponement of the treatment is left to the discretion of the PI.

  ** Women of non-childbearing potential:
  1. At least 12 months since the last menses, or
  2. Without uterus and/or both ovaries, or
  3. Has been surgically sterile for at least 6 months prior to trial drug administration.

     * Acceptable methods of birth control which are considered to have a low failure rate (i.e., less than 1% per year) when used consistently and correctly, such as implants, injectable, combined (estrogen/progesterone) oral contraceptives, intrauterine devices (IUDs-only hormonal), condoms with spermicide, sexual abstinence or vasectomized partner.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2028-04-01 (Estimated); Study Completion 2029-04-01 (Estimated)

PRIMARY OUTCOMES:
Complete Response (CR) Rate | At the end of the initial 6-week induction phase (up to 12 weeks if re-induction is necessary)
  The proportion of participants who achieve a complete response, defined as the absence of detectable high-grade disease via ureteroscopy, imaging (CTU/MRU), and urine cytology following the completion of the initial Gem/Jel treatment regimen. A complete response indicates no visible tumor during endoscopic evaluation and no evidence of cancer cells in collected samples

SECONDARY OUTCOMES:
Safety and Incidence of Adverse Events | Throughout the study period (up to 3 years)
  Frequency and severity of adverse events associated with the sequential Gem/Jel treatment, including drug-related toxicities and complications related to the nephrostomy tube, evaluated using Common Terminology Criteria for Adverse Events (CTCAE) criteria CTCAE) guidelines, which categorize the severity of side effects on a scale from mild (grade 1) to severe (grade 5).

IPD SHARING:
Plan to Share IPD: No